CLINICAL TRIAL: NCT05556122
Title: Efficacy of Compound Betamethasone Injection Combined With Ropivacaine in Ultrasound-guided Slit Intercostals Nerve Block for Chronic Post-thoracotomy Pain:A Single Blind Randomized Control Trial
Brief Title: Efficacy of Compound Betamethasone Injection Combined With Ropivacaine in Ultrasound-guided Intercostal Nerve Block for Chronic Post-thoracotomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yibin Qin, associate chief physician, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-K107-01
Record Dates: First submitted 2022-09-19; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Nerve Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intercostal nerve block at the incision (Experimental): General anesthesia and intercostal nerve block were performed.The drug for intercostal nerve block was 0.33% ropivacaine +2.333mg compound betamethasone (1.667mg betamethasone dipropionate + 0.667mg betamethasone sodium phosphate) to 15ml
  Interventions: Other: intercostal nerve block; Drug: ropivacaine + compound betamethasone
- lateral intercostal nerve block at costal angle (Active Comparator): General anesthesia and intercostal nerve block were performed.The drug for intercostal nerve block was 0.33% ropivacaine +2.333mg compound betamethasone (1.667mg betamethasone dipropionate + 0.667mg betamethasone sodium phosphate) to 15ml
  Interventions: Other: lateral intercostal nerve block; Drug: ropivacaine + compound betamethasone

INTERVENTIONS:
Other: intercostal nerve block — General anesthesia and intercostal nerve block were performed. The drug for intercostal nerve block was 0.33% ropivacaine +2.333mg compound betamethasone (1.667mg betamethasone dipropionate + 0.667mg betamethasone sodium phosphate) to 15ml
  Arms: intercostal nerve block at the incision
Other: lateral intercostal nerve block — lateral intercostal nerve block
  Arms: lateral intercostal nerve block at costal angle
Drug: ropivacaine + compound betamethasone — The drug for intercostal nerve block was 0.33% ropivacaine +2.333mg compound betamethasone (1.667mg betamethasone dipropionate + 0.667mg betamethasone sodium phosphate) to 15ml

SUMMARY:
The patients were divided into two groups by random number method: GroupRD1 group and GroupRD2 group were given general anesthesia and intercostal nerve block.The drug for intercostal nerve block was 0.33% ropivacaine +2.333mg compound betamethasone (1.667mg betamethasone dipropionate + 0.667mg betamethasone sodium phosphate) to 15ml.

DETAILED DESCRIPTION:
The RD1 group received ultrasound-guided intercostal nerve block at the incision before anesthesia induction, and the RD2 group received ultrasound-guided intercostal nerve block at the lateral costal Angle before anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old
2. ASA grade I-III
3. BMI: 18.5-28kg/m2
4. Type of surgery: elective thoracoscopic lung mass resection
5. Informed consent has been signed by the patient and/or family members

Exclusion Criteria:

1. game anesthesia or sugar cortical hormone drugs allergic
2. preoperative use of opioid medicines
3. serious blood coagulation dysfunction
4. serious heart, lung, liver and renal insufficiency
5. put, chemotherapy, and glucocorticoid immunosuppressive therapy history or diseases of the immune system
6. peptic ulcer
7. newly gastrointestinal surgery
8. has a history of thoracic surgery
9. is the central nervous system disease
10. Other glucocorticoids should be used with caution in patients such as fractures, wound repair, corneal ulcers, hyperadrenocortical disease, diabetes mellitus, pregnant women, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute and chronic postoperative pain | 6 hours after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain
Acute and chronic postoperative pain | 24 hours after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain
Acute and chronic postoperative pain | 48 hours after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain
Acute and chronic postoperative pain | 1 months after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain
Acute and chronic postoperative pain | 3 months after surgery
  Numeric rating scale(NRS) is used to assess acute postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: DingYing Ge, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- YiBinQin, Nantong, Jiangsu, China